CLINICAL TRIAL: NCT05775705
Title: The Efficacy and Safety of L-DEP Regimen Combined With PD-1 Antibody an Induction Therapy for Epstein-Barr Virus (EBV)-Positive Lymphoma-associated Hemophagocytic Lymphohistiocytosis
Brief Title: L-DEP Regimen Combined With PD-1 Antibody as Induction Therapy for Epstein-Barr Virus-positive LA-HLH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Professor and Head of hematology, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH20220920001
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: PD-1 Antibody; Hemophagocytic Lymphohistiocytosis; Epstein-Barr Virus; Lymphoma
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Epstein-Barr Virus Infections; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-DEP and PD-1 antibody (Experimental): PEG-aspargase, liposomal doxorubicin, etoposide, and methylprednisolone administered in 2 week cycles for 2 cycles
  Interventions: Drug: L-DEP and PD-1 antibody

INTERVENTIONS:
Drug: L-DEP and PD-1 antibody — Doxorubicin (doxorubicin hydrochloride liposome injection) 35 mg/m2 day 1; etoposide 75 mg/m2 day1; methylprednisolone 1.5mg/kg days 1 to 3, 0.25mg/kg day 4 to 14; PEG-aspargase 6000iu/m2 day2, day4; PD-1 antibody injection 200mg day 5.

SUMMARY:
The efficacy and safety of L-DEP (PEG-aspargase, liposomal doxorubicin, etoposide, and methylprednisolone) regimen combined with PD-1 Antibody an induction therapy for Epstein-Barr virus (EBV)-positive lymphoma-associated hemophagocytic lymphohistiocytosis.

DETAILED DESCRIPTION:
Lymphoma-associated hemophagocytic lympohistiocytosis is a refractory immune disorder with high mortality. Without early intervention, the median survival time is less than 2 months. Currently, HLH-94 or HLH-04 are the standard HLH treatment regimens, which have improved the disease response rate to approximately 70% and increased the 5-year OS rate to 50%. However, approximately, 30% of the patients remain unresponsive to standard therapy, especially if HLH is lymphoma-associated. Therefore, we conduct a prospective clinical study to explore the efficacy and safety of L-DEP (PEG-aspargase, liposomal doxorubicin, etoposide, and methylprednisolone) regimen combined with PD-1 Antibody an induction therapy for Epstein-Barr virus (EBV)-positive lymphoma-associated hemophagocytic lymphohistiocytosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as lymphoma-Hemophagocytic Lymphohistiocytosis.
* EBV-DNA in peripheral blood > 1000 copies/ml or EBER detected in tissue specimens.
* Age 18~65，gender is not limited.
* Estimated survival time ≥ 1 month.
* Cardiac ultrasound LVEF≥50%; No Active bleeding of the internal organs(digestive tract, lung, brain, etc.); If the patient has dyspnea, oxygenation index >250.
* Signed informed consent.

Exclusion Criteria:

* Heart function above grade II (NYHA).
* Severe myocardial injury：TNT、TNI、CK-MB > 3 ULN.
* Accumulated dose of doxorubicin above 400mg/m2 、epirubicin above 750mg/m2、pirarubicin above 800mg/m2 or the patients treated with anthracycline induced cardiovascular disease.
* Pregnancy or lactating Women.
* Allergic to pegylated liposomal doxorubicin，etoposide，or PD-1 antibody.
* Thyroid dysfunction.
* HIV antibody positivity.
* Acute or chronic active hepatitis B (HBsAg positivity, HBV DNA negative acceptable), acute or chronic active hepatitis C (HCV antibody negatively acceptable; HCV antibody positivity, HCV RNA negative acceptable).
* Participate in other clinical research at the same time.
* The researchers considered that patients are not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | Two weeks after initiation of L-DEP regimen combined with PD-1 antibody
  complete response (CR) and partial response (PR) rates

SECONDARY OUTCOMES:
Response rate of lymphoma | Four weeks after second cycle of L-DEP and PD-1 antibody regimen
  complete response (CR) and partial response (PR) rates, using the standard response criteria
Progression Free Survival | 1 years
  from date of inclusion to date of progression, relapse, or death from any cause
Overall Survival | 1 years
  from the date of inclusion to date of death, irrespective of cause
Adverse Events | 30 days after last administration of cytotoxic drugs
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No